CLINICAL TRIAL: NCT04781595
Title: Effect of Watermelon and Beetroot Products on Endothelial Function in Young and Older Adults
Brief Title: Watermelon and Beetroot Products on Endothelial Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Thiago Alvares, Principal Investigator, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: E-26/202.905/2019
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Healthy Young; Older People With Cardiovascular Disease Risk
Keywords: endothelial function; L-citrulline; nitrate; nitric oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Watermelon (Active Comparator): Watermelon powder containing 3 g of L-citrulline.
  Interventions: Dietary Supplement: Watermelon
- Beetroot (Active Comparator): Beetroot powder containing 8 mmol of nitrate.
  Interventions: Dietary Supplement: Beetroot
- Watermelon + beetroot (Active Comparator): Watermelon powder containing 3 g of L-citrulline and Beetroot powder containing 8 mmol of nitrate.
  Interventions: Dietary Supplement: Watermelon + beetroot
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Watermelon — A single dose of watermelon powder containing 3g of L-citrulline
  Arms: Watermelon
Dietary Supplement: Beetroot — A single dose of beetroot powder containing 8 mmol of nitrate
  Arms: Beetroot
Dietary Supplement: Watermelon + beetroot — A single dose of watermelon and beetroot powder containing 3g of L-citrulline and 8 mmol of nitrate
  Arms: Watermelon + beetroot
Dietary Supplement: Placebo — A single dose of maltodextrin
  Arms: Placebo

SUMMARY:
Cardiovascular disease is the main cause of death worldwide. Endothelial dysfunction is the first step to development of cardiovascular diseases. Endothelial dysfunction occurs due to reduction in nitric oxide, a molecule that plays an important role on vascular health. Due to important role of nitric oxide in endothelial function, several studies have evaluated the effect of its precursors, such as L-citrulline and nitrate on endothelial function parameters. The present study will evaluate the effect of L-citrulline and nitrate derived by watermelon and beetroot products, respectively, on endothelial function of young and older participants. Furthermore, we will evaluate the plasmatic amino acids, nitrate, glucose and insulin in response to ingestion of these products.

ELIGIBILITY:
Inclusion Criteria for healthy young participants:

* Age between 18-35 years;
* Triglycerides ≤ 150 mg/dL
* HDL-cholesterol ≥ 50 mg/dL for women and ≥ 40 mg/dL for men;
* Waist circumference ≤ 102 cm for men and ≤ 88 cm for women).

Inclusion Criteria for older people with cardiovascular risk:

* Age ≥ 60 years;
* Elevated triglycerides ≥150 mg/dL;
* Reduced HDL-cholesterol ≤ 50 mg/dL for women and ≤ 40 mg/dL for men;
* Elevated waist circumference ≥102 cm for men and ≥ 88 cm for women).

Exclusion Criteria:

* Elevated fasting glucose (≥100 mg/dL);
* Smoking;
* Beetroot or watermelon allergy;
* Unwillingness to avoid beetroot or watermelon products during the entire study;
* Other chronic diseases (diabetes, liver disease, etc.) or acutely ill

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilation (FMD) | This measure will be evaluate before the nutritional intervention
Flow-mediated dilation (FMD) | This measure will be evaluate 60 minutes after the nutritional intervention
Flow-mediated dilation (FMD) | This measure will be evaluate 120 minutes after the nutritional intervention
Muscle oxygen saturation | This measure will be evaluate before the nutritional intervention
Muscle oxygen saturation | This measure will be evaluate 30 minutes after the nutritional intervention
Muscle oxygen saturation | This measure will be evaluate 60 minutes after the nutritional intervention
Muscle oxygen saturation | This measure will be evaluate 90 minutes after the nutritional intervention
Muscle oxygen saturation | This measure will be evaluate 120 minutes after the nutritional intervention

SECONDARY OUTCOMES:
Plasmatic amino acids | This measure will be evaluate before the nutritional intervention
Plasmatic amino acids | This measure will be evaluate 30 minutes after the nutritional intervention
Plasmatic amino acids | This measure will be evaluate 60 minutes after the nutritional intervention
Plasmatic amino acids | This measure will be evaluate 90 minutes after the nutritional intervention
Plasmatic amino acids | This measure will be evaluate 120 minutes after the nutritional intervention
Plasmatic glucose | This measure will be evaluate before the nutritional intervention
Plasmatic glucose | This measure will be evaluate 30 min after the nutritional intervention
Plasmatic glucose | This measure will be evaluate 60 min after the nutritional intervention
Plasmatic glucose | This measure will be evaluate 90 min after the nutritional intervention
Plasmatic glucose | This measure will be evaluate 120 min after the nutritional intervention
Plasmatic insulin | This measure will be evaluate before the nutritional intervention
Plasmatic insulin | This measure will be evaluate 30 min after the nutritional intervention
Plasmatic insulin | This measure will be evaluate 60 min after the nutritional intervention
Plasmatic insulin | This measure will be evaluate 90 min after the nutritional intervention
Plasmatic insulin | This measure will be evaluate 120 min after the nutritional intervention

CONTACTS AND LOCATIONS:
Overall Officials: Thiago Alvares, PhD, Principal Investigator — Universidade Federal do Rio de Janeiro
Locations (1):
- Universidade Federal do Rio de Janeiro, Macaé, Rio de Janeiro, Brazil

REFERENCES:
- [Derived] Volino-Souza M, Oliveira GV, Tavares AC, Souza K, Alvares T. The effect of microencapsulated watermelon rind (Citrullus lanatus) and beetroot (Beta vulgaris L.) ingestion on ischemia/reperfusion-induced endothelial dysfunction: a randomised clinical trial. Food Funct. 2023 Aug 29;14(17):7959-7968. doi: 10.1039/d3fo02612d. PMID 37561087
- [Derived] Volino-Souza M, de Oliveira GV, Conte-Junior CA, Alvares TS. Effect of microencapsulated watermelon (Citrullus Lanatus) rind on flow-mediated dilation and tissue oxygen saturation of young adults. Eur J Clin Nutr. 2023 Jan;77(1):71-74. doi: 10.1038/s41430-022-01200-8. Epub 2022 Sep 15. PMID 36109652